CLINICAL TRIAL: NCT04130789
Title: Personalized Swiss Sepsis Study: With Machine Learning and Computational Modelling Towards Personalized Sepsis Management - Discovery of Digital Biomarkers
Brief Title: Personalized Swiss Sepsis Study
Acronym: PSSS_digital
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Personalized Health Network (SPHN) (Unknown); Personalized Health and Related Technologies (PHRT) initiative of ETH Zürich (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-01088; qu18Egli2
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Sepsis
Keywords: clinical data warehouse (CDWH); machine learning; data-driven algorithms; multi-dimensional modelling
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with sepsis (cases): patients who developed or were admitted with sepsis to the ICU (cases)
  Interventions: Other: compare data patterns by data-driven algorithms to determine sepsis; Other: compare data patterns by data-driven algorithms to predict sepsis-related mortality
- patients without sepsis (controls): patients who did not develop sepsis (controls).
  Interventions: Other: compare data patterns by data-driven algorithms to determine sepsis; Other: compare data patterns by data-driven algorithms to predict sepsis-related mortality

INTERVENTIONS:
Other: compare data patterns by data-driven algorithms to determine sepsis — compare data patterns by data-driven algorithms including machine learning and multi-dimensional modelling to reliably determine sepsis
Other: compare data patterns by data-driven algorithms to predict sepsis-related mortality — compare data patterns by data-driven algorithms including machine learning and multi-dimensional modelling to to predict sepsis-related mortality

SUMMARY:
This multi-center study is to focus on patients with sepsis in Intensive Care Units (ICUs) in order to better understand the complex host-pathogen interaction and clinical heterogeneity associated with sepsis. Understanding this heterogeneity may allow the development of novel diagnostic approaches. Data from patients will be analyzed using state-of-the art analytical algorithms for biomarker discovery including machine learning and multidimensional mathematical modelling to explore the large datasets generated. In order to discover digital biomarkers for the study endpoints a case-control study design will be used to compare data patterns from patients with sepsis (cases) and those without sepsis (controls).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an ICU on a Swiss University Hospital.
* Patients expected to stay at least 24h on the ICU

Inclusion Criteria (cases)

* Present at admission to ICU or subsequent development of sepsis 3.0 criteria

Inclusion Criteria (controls)

* Patients not fulfilling sepsis definition during the ICU stay

Exclusion Criteria:

* Decline of general consent or any other negative statement against using data for research.
* Patients with a clear elective stay on the ICUs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients on a Swiss University Hospital ICU from 01.08.2019
Sampling Method: Probability Sample
Enrollment: 17500 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
sepsis-related mortality (sensitivity) | time- series data collected from hospital entry until maximum 12 months after hospital exit (no exact time point specified)
  Algorithm to predict sepsis-related mortality (sensitivity)
sepsis-related mortality (specificity) | time- series data collected from hospital entry until maximum 12 months after hospital exit (no exact time point specified)
  Algorithm to predict sepsis-related mortality (specificity)
Determination of sepsis | time- series data collected from hospital entry until hospital exit; an average of 1 month (no exact time point specified)
  Algorithm to determine sepsis at an early stage (at least 12 hours before classical definitions)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, PD Dr., Principal Investigator — Clinical Microbiology, University Hospital Basel
Locations (16):
- Switzerland (16):
  - Clinical Microbiology, University Hospital Basel, Basel
  - Infectious Diseases and Hospital Epidemiology, University Hospital Basel, Basel
  - Medical Intensive Care Unit; University Hospital Basel, Basel
  - Surgical Intensive Care Unit, University Hospital Basel, Basel
  - Institute for Infectious Diseases, University of Bern, Bern
  - Division Infectious Diseases, University Hospital Bern, Bern
  - Intensive Care Medicine, University Hospital Bern, Bern
  - Division Bacteriology Laboratory, University Hospital Geneva, Geneva
  - Division Infectious Diseases, University Hospital Geneva, Geneva
  - Intensive Care Medicine, University Hospital Geneva, Geneva
  - Division Intensive Care Medicine, University Hospital Lausanne, Lausanne
  - Institute of Microbiology, University Hospital Lausanne, Lausanne
  - Service Infectious Diseases, University Hospital Lausanne, Lausanne
  - Institute for Medical Microbiology, University Hospital Zurich, Zurich
  - Division Infectious Diseases, University Hospital Zurich, Zurich
  - Institute for Intensive Medicine, University Hospital Zurich, Zurich